CLINICAL TRIAL: NCT02221609
Title: Movement System Impairment Based Classification Versus General Exercise for Chronic Non-specific Low Back Pain: a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Pontifícia Universidade Católica de Minas Gerais (Other)
Responsible Party: Principal Investigator, Daniel Camara Azevedo, Phd candidate, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17660913.0.0000.5137
Record Dates: First submitted 2014-08-16; First posted 2014-08-20 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Low Back Pain
Keywords: Low Back Pain, Mechanical Low Back Pain, Low Back Ache, Low Backache, Lower Back Pain, Lumbago
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment based on Movement System Impairment based model (Experimental): Treatment based on Movement System Impairment based classification model is composed by patient education, analysis and modification of daily living activities and prescription of specific exercises
  Interventions: Other: Treatment based on Movement System Impairment model
- General exercise (Active Comparator): The general exercise program consists of stretching exercises of the trunk and lower limbs muscles and strengthening exercises of the trunk muscles (Hayden et al., 2005; Rainville et al., 2004).
  Interventions: Other: General exercise

INTERVENTIONS:
Other: Treatment based on Movement System Impairment model — The analysis and modification of daily activities will be performed by identifying and analyzing the patients activities that provoke their symptoms. The patient will be taught on how to correct his posture and limit the movements that increase the amount of stress on the lumbar spine. The prescription of specific exercises is done based on the patient's classification into one of 5 categories of the MSI model. These exercises consist of practicing the movement tests performed at the initial assessment in a corrected form, emphasizing the control of the lumbar spine movement and increasing movement on the adjacent joints. Patients will also advised to repeat the exercises at home at least once a day. 12 treatment sessions are planned for each patient (2 sessions per week during the first 4 weeks and 1 session per week during the last 4 weeks). Each treatment session has an estimated duration of 45-60 minutes. Patients will register their home exercise in an exercise diary.
  Arms: Treatment based on Movement System Impairment based model
Other: General exercise — The general exercise program consists of 12 treatment sessions with estimated duration between 45-60 minutes per session (2 sessions per week for the first 4 weeks and 1 session per week in last 4 weeks). Each session is also done individually by a trained physical therapist. The patients perform an exercise program that starts with a 5-minutes warm-up followed by stretching exercises. Those stretching exercises address the six directions of lumbar motion and the lower limbs muscles. The patient also performs strengthening exercises of the trunk muscles. Based on correct performance of the exercises, the subject may progress through increased load as tolerated. He is also advised to perform these exercises at home and receive figures of the exercises with written instructions. The exercise program will be adapted according to American College of Sports Medicine recommendations (Garber et al., 2011). Patients will register their home exercise in an exercise diary.
  Arms: General exercise

SUMMARY:
The objective of this study is to investigate the efficacy of a treatment based on Movement System Impairment based classification (MSI) model in patients with chronic non-specific low back pain.

DETAILED DESCRIPTION:
The subjects will be recruited from orthopedic outpatient clinics as well from the community. The examiner will screen the eligibility of each subject based on the eligibility criteria. All eligible subjects will receive information about the study and will sign an informed consent form before participating in the study.

The examiner will collect the baseline data prior to randomisation. This examiner will be blinded to patients' allocation to treatment groups. The subjects will be randomly allocated to one of two groups (treatment based on MSI model or general exercise) using a computer-generated randomisation schedule conducted by a study researcher who will not be involved with the patients and assessment of outcomes. Participant allocation will be kept in a sealed opaque envelopes using a random numerical sequence. The examiner, responsible for the treatment will open the envelope in front of the patient and will communicate him about which treatment group he will be part of. The clinical outcomes of this study will be assessed before, after the treatment (2 months) and at 4 and 6 months after randomisation.

Descriptive analyses will be done to check for data normality. The between-group comparisons to obtain the mean effects of the treatments will be conducted by means of interaction terms (group versus time interactions) using Linear Mixed Models. All data will be given to a statistician who will perform the statistical analysis in coded form. The statistical analysis will be done according to the principles of intention to treat. The SPSS 19 and SigmaPlot 10 will be used for these analyses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both genders between 18 and 65 years of age with chronic non-specific LBP (pain for more than 3 months) with a pain intensity of at least 3 points measured by a 0-10 points pain numerical rating scale
* Subjects must be able to stand and walk independently
* Subjects must be able to read in Portuguese

Exclusion Criteria:

* Subjects with any contraindication to physical exercise according to the guidelines of the American College of Sports Medicine
* Subjects with severe depression (measured by depression, anxiety and stress scale - DASS)
* Subjects with serious spinal pathologies (fractures, tumors, and inflammatory pathologies such as ankylosing spondylitis), nerve root compromise (disc herniation and spondylolisthesis with neurological compromise, spinal stenosis, and others), serious cardiorespiratory diseases, previous back surgery or pregnancy.
* Subjects that cannot be classified into any of the five categories of the Movement System Impairment model upon initial assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 2 months after randomisation
  Pain Intensity will be measured by an 11-point (0-10) Numerical Rating Scale (Pain NRS)
Disability | 2 months after randomisation
  Disability will be measured by the 24-item Roland Morris Disability Questionnaire

SECONDARY OUTCOMES:
Pain Intensity | 4 and 6 months after randomisation
  Pain Intensity will be measured by an 11-point (0-10) Numerical Rating Scale (Pain NRS)
Disability | 4 and 6 months after randomisation
  Disability will be measured by the 24-item Roland Morris Disability Questionnaire
Global perceived effect | 2, 4 and 6 months after randomisation
  Global perceived effect will be measured by an 11-point (-5 to +5) Global Perceived Effect Scale

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Costa, PhD, Principal Investigator — Universidade Cidade de Sao Paulo
Locations (1):
- Pontificia Universidade Catolica de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Hayden JA, van Tulder MW, Malmivaara A, Koes BW. Exercise therapy for treatment of non-specific low back pain. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD000335. doi: 10.1002/14651858.CD000335.pub2. PMID 16034851
- [Background] Rainville J, Hartigan C, Martinez E, Limke J, Jouve C, Finno M. Exercise as a treatment for chronic low back pain. Spine J. 2004 Jan-Feb;4(1):106-15. doi: 10.1016/s1529-9430(03)00174-8. PMID 14749199
- [Derived] Azevedo DC, Ferreira PH, Santos HO, Oliveira DR, Souza JVL, Costa LOP. Baseline characteristics did not identify people with low back pain who respond best to a Movement System Impairment-Based classification treatment. Braz J Phys Ther. 2020 Jul-Aug;24(4):358-364. doi: 10.1016/j.bjpt.2019.05.006. Epub 2019 Jun 13. PMID 31230988
- [Derived] Azevedo DC, Ferreira PH, Santos HO, Oliveira DR, de Souza JVL, Costa LOP. Movement System Impairment-Based Classification Treatment Versus General Exercises for Chronic Low Back Pain: Randomized Controlled Trial. Phys Ther. 2018 Jan 1;98(1):28-39. doi: 10.1093/ptj/pzx094. No abstract available. PMID 29077963